CLINICAL TRIAL: NCT02640183
Title: Lidocaine-Prilocaine (EMLA®) Cream in Hysteroscopy Practice: A Prospective Randomized Non-blinded Controlled Study
Brief Title: EMLA Cream in Hysteroscopy Practice
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Hamdy Bakry Mohye Soliman El Kinawy, TA, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMLA-Hsc
Record Dates: First submitted 2015-12-22; First posted 2015-12-28 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Anesthetics, Local

ARMS (2):
- Group A (EMLA) (Experimental): 3 mL EMLA® cream 5% will be applied in the endocervical canal 7 min before procedure, with a 5-mL needleless syringe. A subsequent application will be made with a swab at ectocervix level, using a vaginal speculum, which will be then withdrawn.
  Interventions: Drug: EMLA
- Group B (Placebo) (Placebo Comparator): 3 mL of ultrasonic gel will be applied in the endocervical canal 7 min before procedure, with a 5-mL needleless syringe. A subsequent application will be made with a swab at ectocervix level, using a vaginal speculum, which will be then withdrawn.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: EMLA
  Arms: Group A (EMLA)
Other: Placebo
  Other Names: Ultrasound gel
  Arms: Group B (Placebo)

SUMMARY:
The aim of this study is to investigate the efficacy of 5% lidocaine 25 mg-prilocaine 25 mg/g cream (EMLA®) applied to the uterine cervix for reducing pain during diagnostic hysteroscopy, using a visual analogue scale (VAS) for pain, and whether it can replace general anesthesia that may be required for some cases of office hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients that must perform a diagnostic hysteroscopy.
2. Acceptance to participate in the study.
3. Signed informed consent.
4. Not taking analgesics (acetaminophen, ibuprofen, mefenamic acid) 6h before admission.
5. Absence of sedative use 24 h before admission

Exclusion Criteria:

1. Hypersensitivity or allergy to anesthetics
2. refusal of the patient
3. Patients under age 18 and pregnant.
4. Patients on anti-arrhythmic drugs due to possibility of drug interaction.
5. Unbearable pain that involves other analgesic measures.
6. Allergic reactions to topical anesthetics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Pain experienced during the procedure scored using a VAS. | Procedure
  All women will be asked to score the pain they experienced during the procedure using a VAS that consists of a 10-cm line scaled from 0 to 10 (0 = no pain and 10 = severe pain). Women will be asked to verbally specify the number that represented their level of perceived pain intensity during the hysteroscopy immediately after the procedure.
  After completing the hysteroscopy, women will be asked if they would recommend the procedure to other women, if they had wished to abandon the hysteroscopy, and whether they would repeat the procedure if needed.